CLINICAL TRIAL: NCT01454960
Title: Use of Behavioral Economics to Improve Treatment of Acute Respiratory Infections (Pilot Study)
Acronym: BEARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Doctor, Associate Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1RC4AG039115-01-2; 1RC4AG039115-01 (NIH)
Record Dates: First submitted 2011-08-04; First posted 2011-10-19 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Acute Respiratory Infections (ARIs)
Keywords: Antibiotics; Inappropriate Prescribing; Respiratory Tract Infections; Behavioral Research
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- SA, AJ, PC (Experimental): Participants are given all 3 interventions:
  Suggested Alternatives, Accountable Justification, and Peer Comparison.
  Interventions: Behavioral: Clinical Decision Support: Accountable Justification; Behavioral: Audit and Feedback: Peer Comparison; Behavioral: CDS Order Sets: Suggested Alternatives
- SA, AJ (Experimental): Participants receive the Suggested Alternatives and Accountable Justification interventions, but not the Peer Comparison intervention.
  Interventions: Behavioral: Clinical Decision Support: Accountable Justification; Behavioral: CDS Order Sets: Suggested Alternatives
- SA, PC (Experimental): Participants receive the Suggested Alternatives and Peer Comparison interventions, but not the Accountable Justification intervention.
  Interventions: Behavioral: Audit and Feedback: Peer Comparison; Behavioral: CDS Order Sets: Suggested Alternatives
- AJ, PC (Experimental): Participants receive the Accountable Justification and Peer Comparison interventions, but not the Suggested Alternatives intervention.
  Interventions: Behavioral: Clinical Decision Support: Accountable Justification; Behavioral: Audit and Feedback: Peer Comparison
- Peer Comparison (Experimental): Participants receive the Peer Comparison intervention, but do not receive the Suggested Alternatives or Accountable Justification interventions.
  Interventions: Behavioral: Audit and Feedback: Peer Comparison
- Suggested Alternatives (Experimental): Participants receive the Suggested Alternatives intervention, but not the Accountable Justification or Peer Comparison interventions.
  Interventions: Behavioral: CDS Order Sets: Suggested Alternatives
- Accountable Justification (Experimental): Participants receive the Accountable Justification intervention, but do not receive the Suggested Alternatives or Peer Comparison interventions.
  Interventions: Behavioral: Clinical Decision Support: Accountable Justification
- Control (No Intervention): Participants do not receive any of the 3 interventions.

INTERVENTIONS:
Behavioral: Clinical Decision Support: Accountable Justification — Accountable Justification is triggered by discordant prescriptions that populate the EHR note with provider's rationale for guideline exceptions (AJ).
  Other Names: AJ; Accountable Justification
  Arms: AJ, PC; Accountable Justification; SA, AJ; SA, AJ, PC
Behavioral: Audit and Feedback: Peer Comparison — Performance feedback that benchmarks providers' own performance to that of their peers (PC, for Peer Comparison).
  Other Names: PC; Peer Comparison
  Arms: AJ, PC; Peer Comparison; SA, AJ, PC; SA, PC
Behavioral: CDS Order Sets: Suggested Alternatives — Order Sets that are triggered by EHR workflow containing exclusively guideline concordant choices (SA, for Suggested Alternatives).
  Other Names: SA; Suggested Alternatives
  Arms: SA, AJ; SA, AJ, PC; SA, PC; Suggested Alternatives

SUMMARY:
Bacteria resistant to antibiotic therapy are a major public health problem. The evolution of multi-drug resistant pathogens may be encouraged by provider prescribing behavior. Inappropriate use of antibiotics for nonbacterial infections and overuse of broad spectrum antibiotics can lead to the development of resistant strains. Though providers are adequately trained to know when antibiotics are and are not comparatively effective, this has not been sufficient to affect critical provider practices.

The intent of this study is to apply behavioral economic theory to reduce the rate of antibiotic prescriptions for acute respiratory diagnoses for which guidelines do not call for antibiotics. Specifically targeted are infections that are likely to be viral.

The objective of this study is to improve provider decisions around treatment of acute respiratory infections.

The participants are practicing attending physicians or advanced practice nurses (i.e. providers) at participating clinics who see acute respiratory infection patients. A maximum of 550 participants will be recruited for this study.

Providers consenting to participate will fill out a baseline questionnaire online. Subsequent to baseline data collection and enrollment, participating clinic sites will be randomized to the study arms, as described below.

There will be a control arm, with clinic sites randomized in a multifactorial design to up to three interventions that leverage the electronic medical record: Order Sets that are triggered by EHR workflow containing exclusively guideline concordant choices (SA, for Suggested Alternatives); Accountable Justification (AJ) triggered by discordant prescriptions that populate the note with provider's rationale for guideline exceptions ; and performance feedback that benchmarks providers' own performance to that of their peers (PC, for Peer Comparison).

The outcomes of interest are antibiotic prescribing patterns, including prescribing rates and changes in prescribing rates over time.

The intervention period will be over one year, with a one-year follow up period to measure persistence of the effect after EHR features are returned to the original state and providers no longer receive email alerts.

DETAILED DESCRIPTION:
Each consented provider will be randomized to 1 of 8 cells in a factorial design with equal probability. If results of retrospective data analysis imply that design will be improved by stratification, randomization will be stratified by factors that could influence outcomes.

Data will be collected from Northwestern University's Enterprise Data Warehouse which houses copies of data recorded in the Epic electronic health record. Data elements from qualifying office visits will be collected from coded portions of the electronic health record.

An encounter is eligible for intervention if the patient's diagnosis is in the selected group of acute respiratory infections. The intervention EHR functions will be triggered when clinicians initiate an antibiotic prescription or enter a diagnosis for an acute respiratory infection that has a defined Order Set. If an antibiotic from a list of frequently misprescribed antibiotics is ordered and a diagnosis has not yet been entered, providers will be prompted to enter a diagnosis. If the diagnosis entered is acute nasopharyngitis; acute laryngeopharyngitis/acute upper respiratory infection; acute bronchitis; bronchitis not specified as acute or chronic; or flu; the interventions will be triggered. The diagnosis-appropriate order set will pop-up for providers in the Suggested Alternatives (SA) arm, while clinicians randomized to the Accountable Justification (AJ) arm will receive an alert and be required to enter a brief statement justifying their antibiotic prescription if antibiotics are not indicated for the diagnosis entered. This note will then be added to the patient's medical record.

Clinicians randomized to the Peer Comparison (PC) condition will receive monthly updates about their antibiotic prescribing practices relative to other clinicians in their practice.

ELIGIBILITY:
Inclusion Criteria:

A practicing attending physician or advanced practice nurse ("provider") at Northwestern University's NMFF GIM Clinic in 2011-2013 who sees acute respiratory infection patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Antibiotic Prescribing Rate for 5 Specific Acute Respiratory Infection Diagnoses | 2 years
  Changes in antibiotic prescribing rate for the following ICD-9 diagnoses:
  460 Acute nasopharyngitis (common cold)
  465 Acute laryngeopharyngitis/acute upper respiratory infection
  466 Acute bronchitis
  490 Bronchitis not specified as acute or chronic
  487 Flu

SECONDARY OUTCOMES:
Antibiotic Prescribing Rates for Expanded List of Acute Respiratory Infection Diagnoses | 2 years
  We will monitor overall prescribing for the specified diagnoses and other Acute Respiratory Infection diagnoses, including cough/fever and pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Persell, MD, Principal Investigator — Northwestern University; Jason N Doctor, PhD, Study Director — University of Southern California
Locations (1):
- Northwestern Medical Faculty Foundation General Internal Medicine Clinic, Chicago, Illinois, United States

REFERENCES:
- [Derived] Persell SD, Doctor JN, Friedberg MW, Meeker D, Friesema E, Cooper A, Haryani A, Gregory DL, Fox CR, Goldstein NJ, Linder JA. Behavioral interventions to reduce inappropriate antibiotic prescribing: a randomized pilot trial. BMC Infect Dis. 2016 Aug 5;16:373. doi: 10.1186/s12879-016-1715-8. PMID 27495917